CLINICAL TRIAL: NCT02307292
Title: Prospective, Non-randomized Post Market Surveillance Registry to Document the Clinical Performance in Routine Clinical Practice of the POLARIS Peripheral Vascular Self Expanding Stent System.
Brief Title: Prospective, Post Market Surveillance Q3-registry (POLARIS)
Acronym: Q3-Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: QualiMed Innovative Medizinprodukte GmbH (Industry)
Responsible Party: Principal Investigator, Hans Krankenberg, MD PhD, Herz- und Gefaesszentrum Bad Bevensen
Other Study IDs: QualiMed
Record Dates: First submitted 2014-11-18; First posted 2014-12-04 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Peripheral Artery Disease
Keywords: Superficial femoral artery; Self Expanding Stent System
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: POLARIS Peripheral Vascular Self Expanding Stent System

SUMMARY:
This is a prospective, non-randomized post market surveillance registry designed to document the clinical Performance in Routine clinical practice of the POLARIS Peripheral Vascular Self Expanding Stent System

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Single target de novo superficial femoral artery lesion (angiographic evidence of >50% Stenosis or occlusion) by visual estimate
* Rutherford category II-IV
* At least one patent outflow artery to the ankle.
* Patient signed the informed consent

Exclusion Criteria:

* Patient with acute or subacute Thrombus
* Patients with hyperkoagulopathy
* Patients with Stenosis or occlusion where lesion crossing with guide wire is not possible
* Pregnancy or positive pregnancy test
* Previous enrolment in this Trial or other industrial Trials
* Patient´s inability to fully cooperate with the registry protocol Patient with cancer Treatment (life expectancy less than 2 years) Patients with renal failure

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with single significant (>50%) superficial femoral artery disease
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Freedom from target lesion revascularization | at 12 months
  Clinically driven

SECONDARY OUTCOMES:
Binary restenosis/ reocclusion | at 12 months
  Defined as peak systolic velocity tatio (PSVR) > 2.4
Target limb amputation at the index leg (major and minor separately) | at 12 months
All-cause death | at 12 months
Change in resting ankle brachial index (ABI) | From baseline to 12 and 24 months
Change in Rutherford Classification | From baseline to 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans Krankenberg, MD,PhD, Principal Investigator — Cardiovascular Center Bad Bevensen, Department of Angiology
Locations (1):
- HGZ Bad Bevensen, Department of Angiology, Bad Bevensen, Germany

REFERENCES:
- [Derived] Thieme M, Arjumand J, Spanagel M, Tepe G, Blessing E, Kroeg B, Reichert V, Betge S, Wickenhofer R, Tessarek J, Ingwersen M, Krankenberg H. Stents With Torsional Strength for Superficial Femoral Artery Disease: The Prospective Q3-Registry. J Endovasc Ther. 2022 Dec;29(6):904-912. doi: 10.1177/15266028211067726. Epub 2022 Jan 7. PMID 34994234